CLINICAL TRIAL: NCT04411498
Title: Effects of Fibromyalgia Syndrome in Patients With Diffuse Systemic Sclerosis: Evaluation With 2010 ACR Criteria Set
Brief Title: Effects of Fibromyalgia Syndrome in Patients With Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Ayan, Principal Investigator, Antalya Training and Research Hospital
Other Study IDs: 2019-041
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Systemic Sclerosis; Fibromyalgia
Keywords: fibromyalgia; systemic sclerosis; quality of life
MeSH Terms: conditions — Scleroderma, Systemic; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of Systemic Sclerosis: Patients who were followed-up with the diagnosis of diffuse systemic sclerosis in the Hospital of Rheumatology Clinic were evaluated in terms of inclusion criteria. 44 female patients who met the inclusion criteria were included in the study. All patients were evaluated by a rheumatologist with detailed history and physical examination. Scleroderma patient group was evaluated for the presence of other rheumatic diseases that may accompany.
  Interventions: Diagnostic Test: Fibromyalgia diagnosis in patients with SSc
- Group of control: The healthy control group (96 female ) was evaluated for rheumatic diseases [undiagnosed connective tissue diseases and additional rheumatological diseases] that may accompany secondary FMS exclusion.
  Interventions: Diagnostic Test: Fibromyalgia diagnosis in patients with SSc

INTERVENTIONS:
Diagnostic Test: Fibromyalgia diagnosis in patients with SSc — American College of Rheumatology (ACR) FMS diagnostic criteria set:It is evaluated by the common pain index [WPI] and symptom severity (SS) scale [19]. Diffuse pain index [WPI]; It is a scale that can be scored between 0-19 and obtained by indicating the aching regions of the patient during the last 1 week. Right shoulder, left shoulder, right hip [gluteal region], left hip [gluteal region], left chin, right chin, left upper arm, left lower arm, right upper arm, right lower arm, left upper leg, left lower leg, includes right upper leg, right lower leg, chest, neck, abdomen, upper back, lower back. Symptom Severity Scale [SSS]; evaluates weakness, tired awakening and cognitive functions. In addition, muscle pain, weakness, irritable bowel syndrome, memory problems, headache, abdominal pain, numbness, dizziness, insomnia, depression, constipation, irritability, dry mouth etc. It also evaluates somatic symptoms.

SUMMARY:
Systemic sclerosis [SSc]; is a multisystem disease characterized by immune activation, microvascular disease and fibroblast dysfunction, which is thought to occur as a result of complex and not fully understood interaction between genetic and environmental factors, leading to fibrotic changes in the skin and some internal organs. It is characterized by the deposition of collagen and other matrix components in the skin and some internal organs. It has been shown by evaluating the health assessment questionnaire that it causes disability with increasing frequency over time.

Although pain cannot be localized too well to be attributed to a particular anatomical area, there are several musculoskeletal pain syndromes that can be detected in patients with systemic sclerosis. These are tendonitis, polyarthritis, rheumatoid arthritis, bursitis and fibromyalgia. While there are several studies on others, the relationship between fibromyalgia syndrome and SSc is not known clearly. As with other connective tissue diseases, fibromyalgia is not considered to be rare in SSc.

DETAILED DESCRIPTION:
There are a few studies on this subject. Except for one of these studies, the sensitive point in ACR 1990 FMS diagnostic criteria set was evaluated. In 2010, ACR published new criteria, which may be an alternative method in clinical practice, without sensitive points, including the common pain index and symptom severity scale. It is evaluated with the common pain index and symptom severity scale. This new set of criteria alone is not affected by pain, it is based on patient reporting. Therefore, it seems clinically more significant in determining the origin of pain in autoimmune diseases. There was only one study in the literature in which SSc patients are evaluated with the 2010 FMS criteria set . Therefore, the aim of our study was to evaluate the frequency of FMS according to 2010 FMS criteria and to investigate its effect on quality of life in our study.

ELIGIBILITY:
Inclusion Criteria:

* SSc diagnosis is definitive and diffuse involvement
* no additional disease known other than scleroderma (Diabetes mellitus, hypertension etc.)
* no known additional rheumatic diseases

Exclusion Criteria:

* To have depression and / or any psychiatric illness
* To use steroid, antidepressant, antiepileptic, regular NSAID usage.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with systemic sclerosis
Study Population: Systemic Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 1 week
  The Fibromyalgia Impact Questionnaire [FIQR] was used to evaluate patients' functional status, disease progression, and outcomes. The Turkish validity study Sarmer et al. This questionnaire consists of 20 questions that question physical function, work status, depression, anxiety, sleep, pain, stiffness, fatigue and well-being. Item 1 is scored between 0-3. Other items range from 0-10 points.The total score ranges from 0-80. 80 points indicate high effectiveness.
Beck anxiety inventory | 1 week
  It was developed by Beck et al. in 1988. It is a scale that measures the severity of anxiety symptoms experienced by individuals and is filled by the patient. Questions subjective subjective anxiety and physical symptoms. It consists of 21 items and it is scored between 0 and 3 likert type. The high scores in the scale indicate the severity of the anxiety experienced by the individual. Turkish validity and reliability study was made by Ulusoy et al.
Beck Depression Inventory | 1 week
  It assesses risk for depression as well as level and changes in severity of depressive symptoms in the patients. This scale was developed by Beck et al. in 1961. BDI is self-reported assessment scale including 21 self-assessment statements which are rated by using 4-points Likert scale. Turkish validity and reliability was proven

SECONDARY OUTCOMES:
Short Form-36 | 1 week
  It is a scale developed to measure the quality of life. Its validity and reliability in Turkish has been made. The SF-36 includes a health transition item and assesses 4 physical healthdomains as well as 4 mental health domains. The SF-36 scales can be summarized into physical component summary [PCS] and mental component summary (MCS)scores. Each SF-36 scale is scored 0-100, a higher score representing better health

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Ethics Commitee of Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is a data (Statistical Package for the Social Sciences-SPSS) to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Perrot S, Peixoto M, Dieude P, Hachulla E, Avouac J, Ottaviani S, Allanore Y. Patient phenotypes in fibromyalgia comorbid with systemic sclerosis or rheumatoid arthritis: influence of diagnostic and screening tests. Screening with the FiRST questionnaire, diagnosis with the ACR 1990 and revised ACR 2010 criteria. Clin Exp Rheumatol. 2017 May-Jun;35 Suppl 105(3):35-42. Epub 2017 Feb 8. PMID 28229811